CLINICAL TRIAL: NCT04365504
Title: Efficacy of Cone Beam Computed Tomography Derived Radiomorphometric Indices in Screening of Post-Menopausal Females for Osteoporosis.
Brief Title: Efficacy of Cone Beam Computed Tomography in Diagnosing Osteoporosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Other Study IDs: HarshaPopli
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Post menopausal females; Cone beam computed tomography
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Osteoporotic: Post menopausal females with Lumbar T score <-2.5 as determined by dual energy X ray absorbitometry
  Interventions: Diagnostic Test: Dual energy X ray absorbtiometry
- Osteopenic: Post menopausal females with Lumbar T score -1 to -2.5 as determined by dual energy X ray absorbitometry
  Interventions: Diagnostic Test: Dual energy X ray absorbtiometry
- Normal: Post menopausal females with T score >-1 as determined by dual energy X ray absorbitometry
  Interventions: Diagnostic Test: Dual energy X ray absorbtiometry

INTERVENTIONS:
Diagnostic Test: Dual energy X ray absorbtiometry — The primary clinical application of dual-energy x-ray absorptiometry (DXA or DEXA) is the measurement of bone mineral content (BMC, g) and bone mineral density (BMD, g/cm2) of the lumbar spine and proximal femur to assess risk for osteoporosis.

SUMMARY:
SUMMARY TITLE: "Efficacy of Cone Beam Computed Tomography derived radiomorphometric indices in screening of postmenopausal females for osteoporosis." RATIONALE: Osteoporosis is a disease of altered bone architecture affecting primarily elderly and middle-aged women and men, particularly post-menopausal women. It is responsible for a high number of fractures and poses a high financial burden in both developed and developing countries. In India, we are in a situation where an important, high- burden disease-osteoporosis is being neglected due to lack of facilities of detection, and unawareness about the other tools of assessing bone mineral density and fracture risk.

Few researchers have explored the use of radiomorphometric indices of Cone Beam Computed Tomography (CBCT) and have concluded that these can be used to differentiate between osteoporotic and non-osteoporotic patients. Increasing use of CBCT for various dental conditions, especially implant planning in older age group of patients, which is prone to osteoporosis, calls for the need for further exploration in this regard. The studies available in the literature are heterogenous in nature and reproducibility of the indices used has not been measured. Also, the sample size in each study was limited alongwith presence of selection bias. Thus, the present study will aim at assessing the efficacy of these indices in CBCT in an Indian population, the studies of which are sparse in literature, which shall aid in timely detection and therefore timely intervention to increase the quality of life and reduce morbidity and mortality occurring as a consequence of this disease.

RESEARCH QUESTION:

P: Population (Postmenopausal females with Osteoporosis i.e. DXA values below -2.5) I: Intervention (none) C: Control (Non-osteoporotic post-menopausal females) O: Outcome (CTCI, CTMI, CTI(S)and CTI(I) scores) T: Time Frame (1 year) S: Study Design (Cross sectional observational study) Setting in Haryana, India

Are radiomorphometric indices of CBCT useful for detecting the presence of postmenopausal osteoporosis?

DETAILED DESCRIPTION:
Osteoporosis is a major health problem worldwide characterized by reduced bone mass and disrupted bone architecture that leads to increased susceptibility to fractures. It has become one of the leading causes of morbidity and mortality in older males and females, occurring more commonly in post-menopausal women.1 The prevalence of osteoporosis varies from 16% to 30% in Caucasian women with 39.7% women risked at sustaining a fracture once in a lifetime.1In a study conducted upon middle aged Indian women, a high prevalence of osteopenia (52%) and osteoporosis (29%) was found, with nutritional deficiency being the causative factor. 2 With such high prevalence rates, the need for timely detection cannot be overemphasized. The disease being largely asymptomatic, comes under the radar of the clinician only when a fracture occurs. The diagnosis is largely centered around measurement of bone mineral density by use of Single and dual X-ray absorptiometry (DXA), Ultrasonic measurement of bone, Computed tomography and Radiography with DXA being the gold standard and also the most commonly used technique.3 Dental radiographs are usually advised for a variety of dental diseases and conditions. This provides an opportunity to use dental radiographs as a screening tool for predicting osteoporosis. The role of pantomographs as a screening tool is well established.8,9 Cone beam computed tomography (CBCT), since its advent in 1999, has been specialised for dental use with its various advantages over conventional CT such as lower exposure dose, higher spatial resolution and space saving. Nowadays, CBCT is the modality of choice for patients requiring implant planning.it provides high resolution images in all three planes thereby allowing accurate quantitative measurements of hard structure. Over the recent years, many clinicians have attempted to establish CBCT as a modality to evaluate bone mineral content(BMC) and have concluded that lumbar vertebrae and femoral neck osteoporosis can be predicted accurately from the radiodensity values of the body of the mandible and it is possible to evaluate BMC from the voxel values of CBCT for dental implant treatment5,6.

However, there is still a controversy regarding use of CBCT for determination of bone quality. CBCT gray values give an approximate density and therefore cannot be expressed as HU as in conventional CT.

Few researchers have explored the use of radio morphometric indices such as computed tomography mandibular index superior (CTI(S)), computed tomography mandibular index inferior (CTI(I)), computed tomography cortical index (CTCI) and the computed tomography mental index (CTMI: inferior cortical width) and have been instrumental in establishing the fact that these indices can be used to differentiate between osteoporotic and non-osteoporotic patients7. Very few studies have been done using CBCT and no such study is available in the literature on an Indian population. Thus, this study will aim at determining the utility of these CBCT indices in detection of osteoporosis (confirmed through DXA scan) to aid in timely detection and therefore timely intervention to increase the quality of life and reduce morbidity and mortality occurring as a consequence of this disease.

ELIGIBILITY:
Inclusion Criteria:

1. Post-menopausal females with atleast 5 years since menopause.
2. Patients undergoing CBCT and DXA within a span of 2 weeks.

Exclusion Criteria:

1. Patients in which pathology is detected at the site of measurements, hindering the calculation of indices.
2. Patients undergoing hormone replacement therapy.
3. Patients with history of diseases affecting bone density- diabetes, thyroid disease, osteoarthritis etc.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Post menopausal females with atleast 5 years since osteoporosis
Study Population: Post-menopausal female patients visiting the Department of Oral medicine and Radiology for CBCT for any dental condition and fulfilling the inclusion criteria will be sent for a DXA scan to measure their bone mineral density. Based on their T scores, 3 groups shall be formed - Osteoporotic, Osteopenic and normal females consisting of a minimum of 16 patients in each group.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2020-02-24 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Radiomorphometric indices of Cone beam computed tomography | one year
  CTCI(CT cortical index) CTMI(CT mental index) CTI(I)(CT mandibular index inferior) CTI(S)(CT mandibular index superior) values

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India